CLINICAL TRIAL: NCT03786679
Title: Non-operative Treatment in Sweden of Proximal Humeral Fratures, a Randomised Multicenter Trial.
Brief Title: Non-operative Treatment in Sweden of Proximal Humeral Fractures
Acronym: NOSWEPH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lars Adolfsson (Other Government)
Responsible Party: Sponsor-Investigator, Lars Adolfsson, Professor, Linkoeping University
Organization: Linkoeping University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06000836
Record Dates: First submitted 2018-11-05; First posted 2018-12-26 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Proximal Humeral Fracture
Keywords: Non-operative treatment, orthosis, healing, rehabilitation
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Outcomes Assessor
Masking Description: The assessors are not involved in the treatment and the radiological assessment of images will be assessed with anonymyized images.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthosis group (Active Comparator): An orthosis with the broken arm in neutral position fixed for four weeks. After these four weeks the patient is instructed to start rehabilitation.
  Interventions: Device: Ultrasling ER III orthosis
- Early rehabilitation group (Active Comparator): The patient is instructed to start early rehabilitation about one week after the trauma.
  Interventions: Device: Ultrasling ER III orthosis

INTERVENTIONS:
Device: Ultrasling ER III orthosis — Application of orthosis and start of rehabilitation after four weeks.

SUMMARY:
Proximal humeral fractures are common especially in the elderly population. The majority of these fractures are minimally displaced and may be treated non-operatively. There is however a controversy about which fractures that need surgery and randomised trials have not been able to show a clinically important advantage in patient reported outcome measures for those operated. The trend is therefore that also displaced and comminute fractures are treated non-operatively. There is however very little scientific support for how the non-operative treatment should be designed and performed. Therefore this prospective multicenter study is aiming at investigating the benefit of a four week immobilisation orthosis as compared to early range of motion exercises for those patients not assigned for surgery one week after the trauma.

ELIGIBILITY:
Inclusion Criteria:

* A proximal humeral fracture verified on radiology no older than 7-10 days.

Exclusion Criteria:

* Surgically treated proximal humeral fracture
* Fracture only involving the greater tuberosity
* Previous surgery in the fractured shoulder
* Ongoing malignancy in the fractured shoulder
* Neurologic disease
* Radiating pain from the neck in the affected arm
* Associated vascular or nerve injuries
* Dementia
* Alcohol abuse
* Unwilling to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2024-02-25 (Estimated); Study Completion 2024-02-25 (Estimated)

PRIMARY OUTCOMES:
Union of fracture | Followed 12 months
  recording of fracture union on radiological images

SECONDARY OUTCOMES:
Oxford shoulder score | 12 months
  Shoulder specific patient reported outcome measure, PROM, with a maximum score of 48 points
Numerical pain reporting scale | 12 months
  Patient reported outcome measure of pain at rest, at night and during activity in scales with 10 steps grading subjective assessment of pain
Quick DASH | 12 months
  Patient reported outcome measure of shoulder function in a 11-item PROM
Global assessment of improvement | 12 months
  Patient rated assessment of global improvement in a numeric scale with 7 steps
Shoulder range of motion | 12 months
  The elevation, abduction, internal and external rotation of the injured shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Lars E Adolfsson, Professor, Principal Investigator — Linkoeping University; Hanna C Björnsson Hallgren, MD, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Lars Adolfsson, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196